CLINICAL TRIAL: NCT00658801
Title: A Phase II Study of Respiratory Gated Proton Beam Radiotherapy for Inoperable Pancreas Carcinoma
Brief Title: Study of Respiratory Gated Proton Beam Radiotherapy for Inoperable Pancreas Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: difficult to register
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Tae Hyun Kim, National Cancer Center Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-07-226
Record Dates: First submitted 2008-03-24; First posted 2008-04-15 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

INTERVENTIONS:
Radiation: Respiratory gated proton beam radiotherapy — Prescription dose to PTV as according to the following dose escalation schema:
  1. Group 1: Tumor size ≤5cm Dose level 1: 60 GyE /20 fx, 3GyE fraction dose, 5 days/week. Dose level 2: 66 GyE /22 fx, 3GyE fraction dose, 5 days/week. Dose level 3: 72 GyE /24 fx, 3GyE fraction dose, 5 days/week.
  2. Group 2: 5cm <Tumor size ≤10cm Dose level 1: 54 GyE /18 fx, 3GyE fraction dose, 5 days/week. Dose level 2: 60 GyE /20 fx, 3GyE fraction dose, 5 days/week. Dose level 3: 66 GyE /22 fx, 3GyE fraction dose, 5 days/week.

SUMMARY:
The only curative option for pancreatic cancer patients is surgery, but the patients within 20% of them are possible for a radical surgery. Accordingly, concurrent chemo-radiation therapy is generally used for palliation of unresectable pancreatic cancer patients. So far, the use of 5-fluorouracil (5-FU) was the traditional method of chemotherapy. However, these days, oral anti-cancer medicine, capecitabine(Xeloda®), was developed and considered as an alternative medicine of 5-fluorouracil (5-FU). Furthermore, according to the recent results of clinical trials, the clinical use of capecitabine(Xeloda®) with radiation therapy was proved to be very effective and safe. Proton therapy is a new radiation therapy which remaining energy is released when they reach the tumor, delivering the most effective dose of radiation and which can minimize the exposure to normal tissues. The purpose of this trial is to improve the therapeutic effects by using proton therapy and chemotherapy concurrently.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed adenocarcinoma of the pancreas or a serum CA19-9 level higher than normal limits and an pancreas cancer-compatible radiological features in one or more in CT/MRI/PET scans
* Unresectable disease base on institutional standard criteria of unresectability or recurrent disease following radical surgery. There is no evidence of metastatic disease in the major viscera and no peritoneal seeding
* Patients with biliary or gastroduodenal obstruction must have drainage prior to starting chemoradiation
* All malignant disease must be encompassable within a single irradiation field (15x15cm maximum)
* All patients must have radiographically assessable disease
* No previous irradiation to the planned field
* Age of ≥ 18 years
* Performance status of 0 to 2 on the Eastern Cooperative Oncology Group (ECOG) score
* Required Entry Labortory Parameters:

  * WBC count ≥ 2,000/mm3
  * hemoglobin level ≥ 7.5 g/dL
  * platelet count ≥ 100,000/mm3
  * total bilirubin ≤ 2.0 mg/dL (Patients with elevated bilirubin due to obstruction should be stented and their bilirubin should be decreased ≤ 2.0 mg/dL prior to study entry)
  * creatinine ≤ 3.0 mg/dL
* Oral intake (including J-tube feeding) of ≥ 1,500 calories/day should be maintained.

Exclusion Criteria:

* There is evidence of metastasis in the major viscera or peritoneal seeding.
* Age of < 18 years
* Previous history of RT adjacent to planned field
* Poor performance status of 3 to 4 on the Eastern Cooperative Oncology Group (ECOG) score
* Pregnant or breast feeding status
* Previous history uncontrolled other malignancies within 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
all cause mortality | two years

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center Korea, Goyang-si, Gyeonggi-do, South Korea